CLINICAL TRIAL: NCT05920057
Title: Effect of Constructive Emotional Management Interventions on Emotional Regulation Difficulties and Peace of Mind Among Older Adults: Current Gap and Future Orientation
Brief Title: Constructive Emotional Management Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rasha salah elsayed eweida, assistant professor, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1512023
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Emotional Regulation; Peace of Mind; Older Adults
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): senior citizens aged 60 and more were randomly assigned into two equal groups at and placed in the study group, which received the constructive emotional management interventions
  Interventions: Behavioral: constructive emotional management interventions
- control group (No Intervention): the control group, which received the elderly clubs' regular services

INTERVENTIONS:
Behavioral: constructive emotional management interventions — The Constructive emotional management interventions sessions were conducted in the activity rooms of the elderly clubs where the researchers met the participants. Participants completed a baseline evaluation of the outcome measures of the researched variables after being found to be eligible for the current study and indicating their willingness to participate willingly. After explaining the study's objectives to participants, the researchers themselves delivered the Constructive Emotional Management Interventions program, which had been vetted by experts in the field.
  Arms: interventional group

SUMMARY:
Emotional dysregulation is considered a phenotypic finding that has a purported impact on older adults' peace of mind. In this venue, employing constructive emotional management intervention is one of the breakthroughs that has been empirically targeted to restore positive emotional states and strengthen mental clarity in the geriatric population. Aim: to determine the effect of constructive emotional management interventions on emotional regulation difficulties and peace of mind among older adults. Design: The present study adopted a quasi-experimental methodological approach.

DETAILED DESCRIPTION:
Most elderly people are emotionally stable and well-regulated up until the age of 70 to 80. Due to the effects of changes in their personal circumstances, some older people, however, regard their mental and physical deterioration as becoming self-evident before they turn 70. In old age, it's normal to experience things like forced retirement, the death of a spouse, changes in the home, or financial insecurity. In old age, a great variety of emotions are felt (Kunzmann et al., 2022).

Emotion is a psychological and cultural adaptation process that enables each person to respond adaptably and dynamically to environmental changes. Emotions add meaning to life, deepen human connections, teach people about their needs and feelings, and inspire them to take action (Troy et al., 2018). The phenomenon of emotions is complex. A single emotion consists of a cognitive evaluation, a bodily sensation, an intention, a personal sentiment, a motor response, and, frequently, an interpersonal component (Rompilla et al., 2022). Everyone, especially older adults, experience emotions on a regular basis. They face a wide range of emotions throughout any given day, along with their highs and lows. While some of these are manageable, others are more intense and challenging. It's common to experience those emotions occasionally. Yet, if they struggle with emotion management for an extended length of time, it may result in mental health issues and emotional regulation difficulties (McRae & Gross 2020).

A response to emotions that is poorly controlled and does not fall within the parameters of an acceptable emotional reaction is referred to as having problems with emotional regulation. The terms marked mood fluctuation, mood swings, and labile mood are also used to describe emotional regulation difficulties. Anger outbursts, anxiety, sadness, substance misuse, suicidal ideation, self-harm, and other self-destructive behaviors may be displayed by older adults who have trouble controlling their emotions. Negative moods, personality disorders, psychosis, and post- traumatic stress disorder are all strongly predicted by problems with emotional regulation. Over time, this disorder may affect older persons' quality of life, social contacts, and personal relationships (Dunn et al., 2018).

One's life balance can be thrown off by negative emotions, which are harmful. Lower mental health and inner peace are associated with higher levels of internal conflict, violence, and negative feelings and ideas. In fact, negative emotions and thoughts play a significant influence in the peace of mind maladjustment. In later life, especially, there may be a considerable correlation between peace of mind and effective emotion control. The spiritual and wisdom frequently represent a sense of inner harmony and a sense of wholeness and integration of the mind and body. The more inner peace elderly people have, the better off their minds are. As a result, regulating emotions may be a key therapy goal in psychological interventions for older persons (Isaacowitz 2022).

A reduction in the ability to control older adults' emotions might happen suddenly, but it can also happen gradually, slowly, and subtly. Hence, gerontological nurses should evaluate and identify any potential mental and emotional distress related to this crucial transitional aging era. Anxiety, despair, worry, and fear are frequently present throughout this time. Also, gerontological nurses should intervene to teach elders how to effectively control and manage their emotions and build personalized plans for each elder. Also, they should take action to stop older persons from making self- destructive decisions and engaging in behaviors like loneliness, sadness, suicide, denial of treatment, and denial of care from family members or medical professionals (Erhan et al.,2021).

Older persons who participate in educational emotional management nursing programs may experience an increase in positive emotions and a decrease in negative ones. The recommended therapies for the current study, constructive emotional management interventions, were constructed on the Dialectical Behavioral Therapy model (DBT). Linehan (2015) developed DBT, a cognitive behavioral treatment that incorporates evidence-based psychotherapy. Borderline personality disorder was its original intended application (BPD). Nowadays, it is utilized to treat a variety of emotional dysregulation and impulse control disorders and symptoms (Linehan & Wilks 2015).

Constructive emotional management therapies, which are based on DBT, are made up of a variety of skills that assist older persons in controlling their emotions, fostering better relationships, and enduring difficult circumstances without impulsivity. These interventions involve skills that should be incorporated and practiced into the daily lives of older individuals. They function similarly to muscles strengthen with use over

time. They instruct elderly people on what best skills are needed, when, and how to implement them. Thus further, constructive emotional management interventions could increase mental clarity, restore emotional dimensions, improve coping mechanisms, and lessen depressive symptoms as people age. The prevention or treatment of mental health issues as well as enhancing mental well-being and peace of mind in old age appear to be potential outcomes of constructive emotional management interventions with an emphasis on emotion-regulation. (Delhom et al., 2018).

ELIGIBILITY:
Inclusion Criteria:1. The ability to write and read. 2. Had a Mini Mental State Examination Scale (MMES) score of 24 or higher, indicating normal cognitive function.

3. Did not have depression, according to the Geriatric Depression Scale Short Form (GDS SF), which has a 0 to 4 score range.

4. Difficulties with emotional regulation: a score of 17 or higher on the Brief Version of the Difficulties in Emotion Regulation Scale: The DERS-16.

-

Exclusion Criteria: those who have cognitive impairment such as dementia

-

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-22 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination Scale (MMES) | 3 month

SECONDARY OUTCOMES:
II) Geriatric Depression Scale- Short Form (GDS-SF) | 3 month

OTHER OUTCOMES:
III) Brief Version of the Difficulties in Emotion Regulation Scale: The DERS-16 | 3 month
IV) The Peace of Mind Scale: PoM | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided